CLINICAL TRIAL: NCT02811029
Title: Language and Motricity in Preterm School Age Children
Acronym: LAMOPRESCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2015/207/HP
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Infant, Premature
Keywords: neurological; difficulties
MeSH Terms: conditions — Premature Birth; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- premature infants less than 32 weeks of age (Experimental): measurement of phonology in premature infants less than 32 weeks of age who participated to LAMOPRESCO-1 study
  Interventions: Behavioral: measurement of phonology

INTERVENTIONS:
Behavioral: measurement of phonology — measurement of phonology will be assess using BILO-3, EDA, VS and VL tests

SUMMARY:
A total of 40% of neurodevelopmental difficulties have been reported in very premature infants less than 32 weeks of age. The Epipage1 study reported a decreasing prevalence of cerebral palsy (9-6%) but a high prevalence of specific cognitive neurological difficulties and an increase in school failure.

Neurocognitive difficulties are numerous: visuospatial dyspraxia, language disorders, executive function disorders as well as attention and behaviour disorders. Developmental language disorders have been rarely reported in the literature. This originally prompted our request i.e. PHRC 2010 National Multicenter: LAMOPRESCO. For the past 3 years this protocol has studied the language development of children who were born very prematurely, aged 3 and a half years free of cerebral palsy, in particular the impact of a short rehabilitation period, precise, at an early stage, and protocolized on a fundamental sensorimotor language. The principal assessment criterion was the measurement of phonology, the cornerstone of oral and written language in humans. The aim of the present project is an analysis of the effect that this specific language stimulation has on the learning of written language. The hypothesis is that a specific work modifying various aspects of a child's language, during the age of 3 to 4, alters the development of phonological skills in a sustainable way. The acquisition of reading skills is basically dependent on the quality of its phonological components. The randomized study of children up to 8 years of age in a cohort of 150 children (LAMOPRESCO) will permit to confirm or refute this hypothesis. These increasing difficulties have been reported as regards the language understanding of 3 to 15 year old children. It is as if the initial difficulties and weaknesses, which moreover constituted oral language, prevented the use or development of neural networks, which became more complex and required both an oral and written language. Are these elements which constitute phonology, at an early stage, modifiable before the close of the clinically measurable developmental window?

ELIGIBILITY:
Inclusion Criteria:

* Randomization in LAMOPRESCO-1 study

Exclusion Criteria:

* None as the same population as in the LAMOPRESCO study will be included

Ages: 8 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of reading speed | Day 1
  Evaluation of reading speed will be assess using silent reading speed test. Patient must read a list of words during 2 minutes. The total number of read words will be analyse to calculate the reading speed.

SECONDARY OUTCOMES:
Evaluation of syntax level | Day 1
  Patient must read a list of words during 2 minutes and select how much words are not correctly written.
Evaluation of vocabulary level, syntax and understanding | Day 1
  Patient must read a list of words during 2 minutes and select how much words are not correctly written.
Evaluation of understanding level | Day 1
  Patient must read a text and then answer oral questions about the history read.

CONTACTS AND LOCATIONS:
Overall Officials: Aude CHAROLLAIS, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No